CLINICAL TRIAL: NCT05674643
Title: Gastric Assessment of Pediatric Patients Undergoing Surgery
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Walid Alrayashi, Director, Regional Analgesia Program, Boston Children's Hospital
Other Study IDs: IRB-P00040829
Record Dates: First submitted 2022-10-18; First posted 2023-01-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Fasting; Delayed Gastric Emptying; Aspiration Pneumonia; Respiratory Aspiration of Gastric Content
Keywords: gastric ultrasound; pre-operative fasting
MeSH Terms: conditions — Fasting; Gastroparesis; Pneumonia, Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - ultrasound and acetaminophen: Cohort 1 will include subjects who have a peripheral intravenous line placed in the pre-op area per routine care. This cohort is on average age 7 years and older. Procedures for cohort 1 will include: (a) gastric US measurement of the antral CSA and gastric volume using the Perlas US qualitative grading assessment by an expert and a novice operator to determine the inter-rater class reliability and repeat measurements by each operator to assess the intra-rater reliability (Aim 1), and (b) serial abdominal ultrasounds for gastric assessment and the acetaminophen absorption test to determine the correlation between gastric US and a gold-standard for gastric emptying (Aim 2). The acetaminophen absorption test requires administering a single weight-based enteral dose of acetaminophen with 6 oz of water and drawing of blood samples through a peripheral intravenous line.
  Interventions: Diagnostic Test: Gastric Ultrasound Baseline Scans; Diagnostic Test: Acetaminophen Absorption Test (AAT); Diagnostic Test: Gastric Ultrasound Serial Scans
- Cohort 2 - ultrasound only: Cohort 2 will include subjects for whom a peripheral intravenous line placement is not part of routine pre-operative care. Average age for cohort 2 is age less than 7 years old. Procedures for Cohort 2 will include a gastric US measurement of the antral CSA and gastric volume using Perlas US qualitative grading assessment by an expert and a novice operator to determine the inter-rater class reliability and repeat measurements by each operator for the intra-rater reliability (Aim 1). This cohort is included to examine the reliability of measurements across age groups.
  Interventions: Diagnostic Test: Gastric Ultrasound Baseline Scans

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound Baseline Scans — The patient's abdomen will be scanned using the ultrasound device by an expert scanner and novice scanner for baseline assessment of the antral CSA and gastric volume using Perlas US qualitative grading assessment.
Diagnostic Test: Acetaminophen Absorption Test (AAT) — Prior to starting the AAT, a baseline plasma acetaminophen level (250 microliters) will be obtained from the intravenous catheter. The subject will then be given 12.5 mg/kg or max 650mg of single batch 32mg/mL acetaminophen followed by 6oz of water PO. Up to 3 additional small volume blood samples will be drawn for acetaminophen levels.
  These additional blood samples (250 microliters each) will be obtained to measure acetaminophen plasma levels at the following goal intervals after acetaminophen administration.T1:10-20 mins, T2:35-45 mins, T3: 60mins. At the time of each lab draw gastric ultrasound will be assessed by the expert scanner to correlate gastric ultrasound with the acetaminophen absorption test as a gold-standard of gastric emptying.
  Groups: Cohort 1 - ultrasound and acetaminophen
Diagnostic Test: Gastric Ultrasound Serial Scans — Cohort 1 will have multiple scans as part of assessing gastric emptying. These sequential scans after the baseline assessment will be done in line with the Acetaminophen Absorption Test timeline (T1:10-20 mins, T2:35-45 mins, T3: 60mins) and will be performed by an expert scanner only.
  Groups: Cohort 1 - ultrasound and acetaminophen

SUMMARY:
The goal of this pilot prospective cohort study is to examine the reproducibility of gastric volume and emptying as measured by gastric ultrasound and its correlation to a gold-standard test for gastric emptying in the perioperative period in pediatric patients. The main questions it aims to answer are:

* What is the reliability (inter-rater variability between expert and novice assessors, and intra-rater variability) of a) the gastric antral cross-sectional area (CSA) and b) gastric volume using the Perlas US qualitative grading assessment, measured by using an ultrasound device in pediatric patients undergoing general anesthesia for elective surgery?
* What is the correlation between ultrasound assessment of gastric emptying by the antral-CSA and gastric emptying determined by the acetaminophen absorption test (AAT), the gold standard?

The study will include two cohorts. Cohort assignment will be based on age and anesthesia induction plan. Subjects >7yrs of age and expected to get an IV induction will be assigned to Cohort #1. Subjects <7yrs of age and not expected to get an IV induction will be assigned to Cohort #2.

* Cohort 1 will include abdominal ultrasound for gastric assessment AND the acetaminophen absorption test which includes administering enteral acetaminophen (tylenol) with 6 oz of water and drawing of blood samples through a peripheral intravenous line.
* Cohort 2 will include subjects for whom a peripheral intravenous line placement is not part of routine pre-operative care. Procedures for Cohort 2 will include abdominal ultrasound only in the pre-op area (no tylenol). This cohort is included to examine the reliability of measurements across age groups.

ELIGIBILITY:
Inclusion Criteria:

* Perioperative patients with ASA classification 1-2
* Ages: 2 years- less than 18 years
* Locations: Longwood and Waltham campuses of Boston Childrens Hospital

Exclusion Criteria:

* History of gastrointestinal surgery
* Gastrostomy
* Known GI dysmotility (cohort 1 only)
* Acetaminophen allergy (cohort 1 only)
* Liver or renal dysfunction- pre-diagnosed or, if available, when serum biomarkers are 2 standard deviations above the highest value considered normal for age. (cohort 1 only)
* Consumption of acetaminophen in the 4 hours prior (cohort 1 only)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study is enrolling healthy pediatric subjects ages 2 through 17 years of age who are undergoing surgery with anesthesia at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability | 1 year
  Measured using the following quantitative and qualitative ultrasound assessments between a novice and an expert gastric ultrasound operator:
  * Qualitative using the previously published Perlas' US qualitative grading assessment
  * Grade 0- no contents visualized in supine and lateral position
  * Grade 1- contents visualized in the lateral decubitus position (RLD) only
  * Grade 2- contents visualized in the supine and RLD.
  * Quantitative assessment using the cross-sectional area as published by Spencer AO et al.
  * Measurement of the CSA: longitudinal diameter (D1), and the antero-posterior diameter (D2) in both supine and RLD. Then these will be used to calculate the cross-sectional area (CSA) = (π*D1*D2)/4.
  * Quantitative assessment using the cross-sectional area as published by Spencer AO et al.
  * Measurement of the CSA: longitudinal diameter (D1), and the antero-posterior diameter (D2) in both supine and RLD. Then these will be used to calculate the cross-sectional area (CSA)
Intra-rater reliability | 1 year
  Measured using the following quantitative and qualitative ultrasound assessments between a novice and an expert gastric ultrasound operator:
  * Qualitative using the previously published Perlas' US qualitative grading assessment
  * Grade 0- no contents visualized in supine and lateral position
  * Grade 1- contents visualized in the lateral decubitus position (RLD) only
  * Grade 2- contents visualized in the supine and RLD.
  * Quantitative assessment using the cross-sectional area as published by Spencer AO et al.
  * Measurement of the CSA: longitudinal diameter (D1), and the antero-posterior diameter (D2) in both supine and RLD. Then these will be used to calculate the cross-sectional area (CSA) = (π*D1*D2)/4.
Gastric Emptying | 1 year
  Outcome will be gastric emptying assessed by the change in antral CSA (measured in cm2) over time after acetaminophen administration, and this will be correlated to gastric emptying over the same period of time by the acetaminophen absorption test PK parameter, AUC60 mcg*min/mL. As such, each patient will act as their own control. Correlation analysis will be applied to examine the performance of CSA measurements overtime using gastric ultrasound to determine gastric emptying compared to the acetaminophen absorption test as the gold standard.

SECONDARY OUTCOMES:
Post-anesthetic outcomes | 1 year
  Fasting times have been correlated to post-anesthetic outcomes such as post-operative nausea/ vomiting, and discomfort, and it is known that some patients fast longer than required by their clinical team, which can result in adverse effects. Reported fasting times for all patients and confirmatory assessment by gastric US will be examined along with data pulled from the medical record about post-operative nausea/ vomiting, post-operative discomfort, satisfaction, and whether the patient met their expected post-operative trajectory or not (e.g. unplanned admission).

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Spencer AO, Walker AM, Yeung AK, Lardner DR, Yee K, Mulvey JM, Perlas A. Ultrasound assessment of gastric volume in the fasted pediatric patient undergoing upper gastrointestinal endoscopy: development of a predictive model using endoscopically suctioned volumes. Paediatr Anaesth. 2015 Mar;25(3):301-8. doi: 10.1111/pan.12581. Epub 2014 Dec 11. PMID 25495405